CLINICAL TRIAL: NCT02091596
Title: Randomized, Double-blind, Vehicle-controlled 2-Arm Trial of Topical PluroGel N for the Treatment of Patients With Mildly Infected Diabetic Foot Ulcer CLINICAL PROTOCOL PGN-1300
Brief Title: Topical PluroGel N for the Treatment of Mildly Infected Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PluroGen Therapeutics, Inc (Industry)
Collaborators: Arkios BioDevelopment International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PGN-1300; D11AC00020 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Foot Ulcer; Infection
Keywords: Wound; Ulcer; Infected; Infection
MeSH Terms: conditions — Diabetic Foot; Infections; Wounds and Injuries; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PluroGel (Placebo Comparator): PluroGel
  Interventions: Drug: PluroGel
- PluroGel N (Experimental): PluroGel N
  Interventions: Drug: PluroGel N

INTERVENTIONS:
Drug: PluroGel N — Study Drug
  Arms: PluroGel N
Drug: PluroGel — PluroGel Vehicle Placebo Comparator
  Arms: PluroGel

SUMMARY:
This will be a randomized, double-blind (evaluator-blind), vehicle-controlled study of 50 enrolled subjects. Adult subjects (greater than 18 years old) who present with a mildly infected diabetic foot ulcer (IDSA criteria) having full thickness (i.e., through the dermis but not involving joint capsule, tendon, and bone). Subjects must also provide informed consent and meet all other entry criteria to be enrolled and randomly assigned to receive PluroGel N or PluroGel vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Non-hospitalized subjects with Type 1 or Type 2 diabetes mellitus as defined by the American Diabetes Association diagnostic criteria (ADA, 2010). Diabetes may be treated with insulin, oral hypoglycemic agents, diet, or a combination of these therapies. Subjects whose diabetes is considered "controlled" by diet or medication in the opinion of the physician.

  * Males or females at least 18 years old.
  * Subjects must be considered by the investigator to be reliable, willing and able to give signed informed consent, and must sign the informed consent form.
  * Subjects must have a full thickness (i.e., extending through dermis but not involving tendon, bone, or joint capsule) ulcer on the foot distal to the malleoli with a surface area ≥1 cm2 after the wound has undergone appropriate debridement. Subjects must have localized mild infection of the ulcer, as defined by the IDSA criteria as per Appendix C, with in the PGN1300 Protocol, which the investigator believes would ordinarily be treated on an outpatient basis.

IDSA mild infection of an ulcer is defined as:

The presence of ≥2 of the following items:

* Local swelling or induration
* Erythema
* Local tenderness or pain
* Local warmth
* Purulent discharge (thick, opaque to white or sanguineous secretion) Local infection involving only the skin and the subcutaneous tissue. If erythema, must be >0.5 cm to ≤2 cm around the ulcer.

  * Diabetic Foot Infection-General Parameters Score of at least 2 must be obtained in order to be eligible for enrollment.
  * Diabetic Foot Infection-Wound Size Score of at least 1 must be obtained in order to be eligible for enrollment.
  * The diagnosis of mild infection must be confirmed immediately following the Day 0 (Enrollment Visit) debridement, although pre-debridement purulence is to be counted as one manifestation of infection.

Exclusion Criteria:

* Subjects with IDSA-defined moderate infection as per Appendix C, including cellulitis extending > 2 cm; lymphangitis; spread beneath the fascia; deep tissue abscess; osteomyelitis; gangrene; muscle, joint, or bone involvement.

  * Subjects with IDSA-defined severe infection as per Appendix C, within PGN1300 Protocol including systemic toxicity or metabolic instability (e.g., fever, chills, tachycardia, hypotension, confusion, vomiting, leukocytosis, acidosis, hyperglycemia, or azotemia).
  * Subjects with systemic inflammatory response signs, as manifested by ≥2 of the following :
* Temperature >38°C or <36°C
* Heart rate >90 beats/min
* Respiratory rate >20 breaths/min or PaCO2 <32 mm Hg
* White blood cell count >12 000 or <4000 cells/μL or ≥10% immature (band) forms

  * Subjects with local wound complications (e.g., prosthetic materials).
  * Subjects currently receiving antibiotic treatment for a localized infection of the study ulcer and whose infection is improving in response to treatment.
  * Subjects requiring concurrent systemic antimicrobials during the study period for any infection, including diabetic foot ulcer.
  * Subjects in whom bone or joint involvement is suspected based on clinical examination (e.g., bone noted visually or by probing) or plain view X-ray.
  * Subjects with clinically significant peripheral arterial disease requiring vascular reconstructive surgery. Subjects who are expected to be unable to care for their ulcer because of hospitalization, vacation, disability, etc. during the study period, or are unable to safely monitor the infection status at home.
  * Subjects with known active alcohol or substance abuse within the 6 months preceding study entry.
  * Subjects who are receiving immunosuppressive agents (other than corticosteroids), radiation therapy, or cytotoxic agents.
  * Subjects who require treatment for a primary or metastatic malignancy (other than squamous or basal cell carcinoma of the skin).
  * Subjects with a systemically immunocompromising disease, such as acquired immune deficiency syndrome or known human immunodeficiency virus infection.
  * Subjects who have had an unexplained fever or chills during the week prior to enrollment.
  * Subjects with other conditions considered by the investigator to be reasons for disqualification that may jeopardize subject safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness, lack of motivation, history of poor compliance).
  * Subjects with any known allergy or other contraindication to any ingredients in the study products.
  * Women who are breast feeding, pregnant, or not using contraception unless sterile.
  * Subjects who have been taking or expect to be taking any other investigational therapy within the 30 days prior to entry or during enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 14 Days
  Clinical Response is defined by the investigator's evaluation of the signs and symptoms of clinical infection.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Ledesma Foot and Ankle, Phoenix, Arizona
  - Foot & Ankle Clinic, Los Angeles, California
  - Samuel Merritt University, Oakland, California
  - ASAP Urgent-Care, Hamden, Connecticut
  - Advance Medical Research Center, Miami, Florida
  - Miami Center for Clinical Research, LLC, Miami, Florida
  - Unlimited Medical Research, LLC, Miami, Florida
  - Phoenix Medical Research, LLC, Miami, Florida
  - Med Research of Florida, LCC, Miami, Florida
  - Sweet Hope Research Specialty, Inc., Miami Lakes, Florida
  - Weil Foot & Ankle Institute, Des Plaines, Illinois
  - Research Integrity, Owensboro, Kentucky
  - Paddington Testing Company, Inc, Philadelphia, Pennsylvania
  - AllCare Foot & Ankle, PA, Arlington, Texas
  - Coastal Podiatry Group, Virginia Beach, Virginia